CLINICAL TRIAL: NCT02451878
Title: Effectiveness and Cost-effectiveness of a Fully Self-guided Internet-based Intervention for Shyness and Sub-clinical Social Anxiety Symptoms in the General Population: Pragmatic Randomised Controlled Trial
Brief Title: Improving Social Anxiety Symptoms (SocWell)
Acronym: SocWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Australian National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MQ14PE_25; Human Ethics Protocol 2015/229 (Other: Australian National University HREC)
Record Dates: First submitted 2015-04-20; First posted 2015-05-22 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2018-07

CONDITIONS: Shyness; Wellbeing
Keywords: shyness; internet; self-help; psychology; wellbeing
MeSH Terms: conditions — Shyness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The E-Couch self-help social anxiety module which is based on cognitive behavioural therapy principles. This module contains a literacy section and 5 toolkits comprising exposure practice, cognitive restructuring (modifying your thinking), attention practice, social skills training and relaxation. E-Couch is designed to be completed at the participant's own pace. It is free to use, browser-based and widely accessible on a range of connected devices.
  Interventions: Behavioral: E-Couch
- Control (No Intervention): Wait list control (WLC)

INTERVENTIONS:
Behavioral: E-Couch — e-couch is an online CBT based intervention
  Arms: Intervention

SUMMARY:
The investigators will test the value of an internet self-help package (E-Couch) for alleviating social anxiety symptoms in the general population. The investigators will undertake a trial of about 2000 participants to compare the effect of the E-Couch intervention compared to a wait-list control condition. Over a period of 12 months the investigators will measure the effect of using E-Couch self-help on social anxiety symptoms, as well as on mental wellbeing, and other secondary outcomes including quality of life, depression and general anxiety, and their use of other sources of help.

DETAILED DESCRIPTION:
DESIGN The study will involve a large, pragmatic, randomised controlled trial of the internet-based self-directed E-Couch social anxiety module versus a wait-list control condition for the reduction of sub-clinical social anxiety symptoms, among a general population sample recruited using direct-to-consumer advertisements on national websites.

RECRUITMENT Participants in this study will be recruited using advertisements placed on websites such as the NHS website. Individuals expressing an interest in the online advertisement by clicking on a web link will be directed to a University website containing full information on the trial and the opportunity to ask questions of the study team by email or telephone. Participants will be advised in the information sheet that they are free to withdraw at any time without giving a reason and without it affecting their care.

CONSENT Interested participants will be asked to indicate their willingness to participate in the screening and/or the trial by clicking on Yes in response to the online consent questions.

SCREENING Users who provide their consent will be invited to complete screening questions which will determine whether they are eligible for participation in the trial.

INCLUSION AND EXCLUSION Inclusion criteria for this trial include age 18 years and over, resident of England and a score of 13 or more on the SPIN social anxiety measure, and a willingness to provide a working email address and mobile phone number (to respond to a confirmation email and receive reminders). People who are currently receiving therapist-guided treatment for social anxiety disorder will be excluded from participation as will those with a self-reported diagnosis of bipolar disorder or schizophrenia.

MEASURES Following completion of the screening survey eligible participants will be advised that they are eligible to participate in the trial and asked to provide their email address and mobile phone number. Once these details have been submitted they will be advised that in 24 hours they will receive an e-mail providing a link to an online baseline survey. The e-mail will link to a battery of demographic and self-report mental health measures. Measures will be taken at baseline and, for those randomised, at all or most of the follow up points including post-intervention, 3-, 6- and 12-months. At each follow-up point both Intervention and Control participants will receive notification of follow-up measures by email and by text message.

RANDOMISATION Participants who complete baseline measures within one week of receiving the survey link via email, will be randomised using an automated computer algorithm to the E-Couch social anxiety tool (Intervention) or to a Wait list control condition. Participants will be advised of the condition to which they have been allocated.

ACCESS TO INTERVENTION Intervention participants will be asked to set a password associated with their email address, and provided with access to the Intervention. Intervention participants will be encouraged to access and use the self-guided intervention over a period of up to 6 weeks (although they can chose to work through the program at their own pace). Access will be via secure login on the research trial website, using their email address and password.

INTERVENTION The E-Couch social anxiety module which is based on cognitive behavioural therapy principles. This module contains a literacy section and 5 toolkits comprising exposure practice, cognitive restructuring (modifying your thinking), attention practice, social skills training and relaxation. E-Couch is designed to be completed at the participant's own pace. It is free to use, browser-based and widely accessible on a range of connected devices.

CONTROL The Control group will be placed on a wait list to receive the intervention in 12 months.

RISKS The risks to the participants are likely to be minimal. The study uses standard well-tested measures or tools modified from these measures. Participants are referred to a source of help in the Information Sheet in case of distress. The intervention has been employed without problems in publically accessible form across the world since 2008.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Resident in England
* Willing to provide email address and mobile telephone number
* Able to use a web-based intervention provided in written English
* SPIN score 13 or more (to include those with subclinical symptoms)

Exclusion Criteria:

* Aged under 18
* Not resident in England
* Unwilling or unable to provide email address and mobile telephone number
* Unable to use a web-based intervention provided in written English
* SPIN score <13
* Self-reported history of psychosis (schizophrenia or bipolar affective disorder)
* Receiving therapist-guided support for social anxiety disorder (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2105 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
change in social anxiety symptoms (self-report using SPIN-17 measure) | change from baseline to 6 weeks
  self-report social anxiety symptoms using SPIN-17 measure

SECONDARY OUTCOMES:
mental wellbeing (self-report WEMWBS measure) | 6 weeks, 3 months, 6 months, 12 months
  mental wellbeing using self-report WEMWBS measure
depression (self-report CES-D measure) | 6 weeks, 3 months, 6 months, 12 months
  depression using self-report CES-D measure
quality of life (using SF36 measure) | 6 weeks, 3 months, 6 months, 12 months
  quality of life using SF36 measure
use of health services (self-reported use of health services)- used for Health economic evaluation. | 12 months
  self-reported use of health services in preceding 3 months
time off work or study (self-reported time off work or study)-Used for health economic evaluation. | 12 months
  self-reported time off work or study in preceding 3 months
social anxiety symptoms (fear of negative evaluation) (self-report using BFNE-S measure) | 6 weeks, 3 months, 6 months, 12 months
  self-report using BFNE-S measure
social anxiety symptoms (self-report using SPIN-17 measure) at secondary time points | 3 months, 6 months, 12 months
  self-report social anxiety symptoms using SPIN-17 measure at secondary time points

CONTACTS AND LOCATIONS:
Overall Officials: John A Powell, PhD, Principal Investigator — University of Oxford; Kathleen M Griffiths, PhD, Principal Investigator — Australian National University
Locations (2):
- National Institute for Mental Health Research, Australian National University, Canberra, Australian Capital Territory, Australia
- Nuffield Department of Primary Care Health Sciences, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Powell J, Williams V, Atherton H, Bennett K, Yang Y, Davoudianfar M, Hellsing A, Martin A, Mollison J, Shanyinde M, Yu LM, Griffiths KM. Effectiveness and Cost-Effectiveness of a Self-Guided Internet Intervention for Social Anxiety Symptoms in a General Population Sample: Randomized Controlled Trial. J Med Internet Res. 2020 Jan 10;22(1):e16804. doi: 10.2196/16804. PMID 31821151
- [Derived] Powell J, Atherton H, Williams V, Martin A, Bennett K, Bennett A, Mollison J, Yu LM, Yang Y, Locock L, Davoudianfar M, Griffiths KM. Effectiveness and cost-effectiveness of a fully self-guided internet-based intervention for sub-clinical social anxiety symptoms: Protocol for a randomised controlled trial. Digit Health. 2017 Apr 10;3:2055207617702272. doi: 10.1177/2055207617702272. eCollection 2017 Jan-Dec. PMID 29942591